CLINICAL TRIAL: NCT07248241
Title: The Caregiver Education Resource for Dementia (CARE-Dem) Study: Developing and Evaluating a Digital Intervention to Support Informal Caregivers of People With Dementia
Brief Title: Developing and Evaluating a Digital Intervention Aiming to Support Informal Caregivers of People With Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Clinical Research and Prevention (Network)
Collaborators: Copenhagen Municipality, Denmark (Other Government); Municipality of Frederiksberg, Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CARE-Dem; J.nr. 2024-0040 (Other Grant/Funding Number: Region Hovedstadens Forskningsfond til Sundhedsforskning)
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-08

CONDITIONS: Dementia Caregiver; Digital Education Interventions
Keywords: Complex Intervention; Intervention Development; Intervention Adaptation; Feasibility; Co-Creation; Informal Caregivers; Support Tool; Digital Intervention; Dementia Caregiving

STUDY DESIGN:
Intervention Model Description: Intervention group receives the intervention, control group receives TAU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants receive the CARE-Dem intervention
  Interventions: Behavioral: Digital support tool
- Control group (No Intervention): Participants receive treatment as usual and can use available offers

INTERVENTIONS:
Behavioral: Digital support tool — The CARE-Dem digital support tool offers a number of modules that participants must complete within three months.
  Arms: Intervention group

SUMMARY:
The goal of this feasibility trial is to test the acceptability and feasibility of a new digital education pro-gram, the Caregiver Education Resource for Dementia (CARE-Dem). This is a behavioral (non-medical) intervention, designed to support informal caregivers of people with dementia. The primary purpose is to explore whether this program can help improve wellbeing and reduce burden among informal caregivers. The study focuses on adult caregivers, such as spouses, partners, relatives, or close friends of people recently diagnosed with dementia or living with mild dementia.

The main questions it aims to answer are:

* Is it possible to recruit and retain caregivers to participate in this type of digital intervention?
* Do participants find the program relevant, useful, and acceptable? Are the study procedures and outcome measures (such as questionnaires) suitable and manage-able for the participants?
* Does the intervention show preliminary signs of reducing caregiver burden and improving care-givers' wellbeing, knowledge, quality of relationship with the person with dementia, ability to ac-cept the situation, and feelings of being capable of managing their caregiving role? Researchers will compare caregivers who receive the CARE-Dem program with a control group who are offered the usual municipal information sessions. This allows us to see whether the digital pro-gram is feasible and whether it shows signs of effect compared with standard practice.

Participants in the intervention group will be asked to:

• Use the CARE-Dem digital platform over a three-month period.

The platform includes three modules:

Module 1: Understanding dementia and medical treatment options Module 2: Everyday life and communication with a person with dementia Module 3: Legal and practical matters, and information on support available in the community

* Engage with a mix of learning materials such as short videos, fact sheets, interactive activities, guides, and links to further resources
* Complete questionnaires at baseline and after 3 months to measure caregiver burden, wellbeing, and self-efficacy
* Take part in qualitative interviews about their experiences with the program, including usability, satisfaction, acquired knowledge, benefits, and suggestions for improvement.

Participants in the control group will receive treatment as usual. They will be offered to take part in existing information sessions provided by the municipalities, but attendance is optional. Researchers will record whether or not they attend, in order to compare results across subgroups.

This feasibility trial will help determine whether it is possible to run a larger evaluation of the CARE-Dem program in the future. If successful, the program could provide flexible and accessible support to the many caregivers of people with dementia, reaching those who cannot attend traditional in-person sessions.

ELIGIBILITY:
Inclusion Criteria:

- Adult family members/relatives/other adult informal caregivers of a newly diagnosed person with dementia/a person with mild dementia

Exclusion Criteria:

* Unable to speak/understand Danish
* Incapable of collaborating about signing the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Baseline minus three months (start of enrollment) to baseline
  Number of participants enrolled divided by number of eligible individuals. Registered by a project nurse at the recruiting clinic
Response rate to survey | Three months (end of intervention)
  Number of full surveys returned at follow-up divided by total number of participants. Assessed in the REDCap database where all survey data are gathered.
User experiences with intervention | Three months (end of intervention)
  Satisfaction, relevance, perceived value, ease of use, key barriers and facilitators for use, suggestions for improvement of the CARE-Dem. Assessed through semi-structured, qualitative interviews with participants in the intervention group.

SECONDARY OUTCOMES:
Barriers to recruitment | Baseline minus three months (start of enrolment) to baseline
  Assessed through semi-structured, qualitative interviews with all professionals involved in re-cruitment and randomisation.
Completeness of survey data | Three months (end of intervention)
  Number of completed survey items at follow-up divided by total number of items. Only surveys filled in at baseline and end of intervention are counted. Assessed in the REDCap database where all survey data are gathered.
Relevance of outcome measures to the target population | Three months (end of intervention)
  Assessed through semi-structured, qualitative interviews with all participants in the intervention group.
Intervention dose received | Three months (end of intervention)
  Proportion of intervention components completed by each participant within three months. Collected via participant logs, where all interaction with the intervention will be documented by participants in the intervention group.
Extent to which the selected outcome measures demonstrate changes in the expected direction and magnitude | Three months (end of intervention)
  Evaluated by comparing observed mean change scores from baseline to end of intervention with effect sizes reported in previous studies of digital interventions for informal caregivers of people with dementia. Feasibility will be considered acceptable if observed changes in the intervention group from baseline to end of intervention are in the expected direction and within the range of small-to-moderate effects (Cohen's d ≥ 0.20), consistent with similar studies of digital interventions for informal caregivers of people with dementia.
Experiences of randomisation procedure | Baseline
  Assessed via short interviews with recruiting nurses who collect accounts from participants in the intervention group and participants in the control group.
Reasons for non-adherence and dropout | Three months (end of intervention)
  Assessed through interviews with participants who do not complete the intervention within the designated three months. We aim to interview as many as possible among participants who drop out or do not complete the intervention.

OTHER OUTCOMES:
Change in caregiver burden from baseline to end of intervention | Baseline and three months
  Measured with the Zarit Burden Interview (ZBI), a 22-item questionnaire including four aspects of caregiver burden: personal strain, role strain, impact on social life, and impact on personal health. Items are rated on a 5-point Likert scale ranging from 0 (never) to 4 (nearly always) with total scores ranging from 0 to 88.
Change in mental wellbeing from baseline to end of intervention | Baseline and three months
  Measured with the World Health Organization 5-Item Well-Being Index (WHO-5), a 5-item ques-tionnaire concerning feelings about everyday life in the previous two weeks. Items are rated on a 6-point Likert scale ranging from 0 (at no time) to 5 (all the time). The raw score ranges from 0 to 25 and is converted to a percentage score from 0 to 100.
Change in self-efficacy from baseline to end of intervention | Baseline and three months
  Measured with the General Self-Efficacy Scale (GSES), a 10-item questionnaire assessing per-ceived ability to cope with challenging and demanding situations. Items are rated on a 4-point Lik-ert scale from 1 (not at all true) to 4 (exactly true) with total scores ranging from 10 to 40.
Acquired knowledge and benefit of the intervention | Three months (end of intervention)
  Participants' experiences of knowledge and benefits acquired from using the intervention, particularly regarding impact on the quality of their relation to the person with dementia, experiences of being able to accept the situation, and feelings of being capable of managing their caregiving role. Assessed through qualitative interviews with participants in the intervention group.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Geriatrics and Palliation, University Hospital Bispebjerg and Frederiksberg ty Hospital, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No